CLINICAL TRIAL: NCT00604097
Title: Preventing Youth Suicide in Primary Care: A Family Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2004-11-3995; 1R49CE000428 (NIH)
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Suicide
Keywords: youth suicide; family therapy; primary care; intervention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Attachment-Based Family Therapy
  Interventions: Behavioral: Attachment-Based Family Therapy
- 2 (Active Comparator): Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Attachment-Based Family Therapy — 12-16 week family-based therapy
  Arms: 1
Behavioral: Enhanced Usual Care — Rapid referral to community outpatient care with weekly monitoring of symptoms by study team
  Arms: 2

SUMMARY:
The purpose of the study is to test the efficacy of a brief family therapy (Attachment-Based Family Therapy) for youth presenting in primary care with suicidal ideation and depressed mood.

DETAILED DESCRIPTION:
Youth suicide is a serious public health problem and clinical challenge for medical and behavioral health providers, yet few preventive interventions have been tested for this population. This project addresses this deficit by testing the efficacy of a brief family therapy for adolescents presenting with serious risk for suicide in a primary care setting. Several innovations characterize the study. First, patients will be identified and treated directly in the primary care setting. Integrating behavioral health services into primary care may a) reduce burden on physicians by promoting parents as safety monitors, b) increase behavioral health treatment adherence, and c) address many underlying family problems associated with suicide. Second, to identify seriously at risk adolescents, we will assess for severe and persistent suicidal ideation and co-occurring depression. Patients will need to score above clinical cutoffs on both ideation (SIQ-JR > 31) and depression (BDI-II >20) at two consecutive appointments (generally within 3 days of each other). Third, treatment will target two of the most critical suicide risk factors: depression and family conflict. Depression is the most consistently associated risk factor for suicide and family conflict is the most common precipitant of completed suicide (20%) and non-fatal suicidal episodes (50%). Fourth, we will use Attachment Based Family Therapy (ABFT; Diamond et al., 2002) as the intervention approach, an efficacious and manualized family therapy model specifically designed for adolescent depression. ABFT has been successful in reducing suicidal ideation, hopelessness, depression, anxiety, and family conflict. Participants will be recruited from the primary care centers at The Children's Hospital of Philadelphia. Eighty-seven percent of patients are African American and 60% are girls. One hundred adolescents will be randomized to 6 to 10 weeks of either ABFT or Enhanced Usual Care (EUC). Patients will be evaluated at baseline 6, 12, 24, and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Suicidal ideation (SIQ-JR > 30)
* Moderate depressed mood (BDI-II > 19)
* At least one parent/caregiver willing to participate

Exclusion Criteria:

* Psychosis
* Mental retardation or other significant cognitive impairment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2004-09; Primary Completion 2007-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation Questionnaire - JR (SIQ-JR) | Baseline, 6 weeks, 12 weels, 24 weeks
Beck Depression Inventory - II (BDI-II) | Baseline, 6 weeks, 12 weeks, 24 weeks
Scale for Suicidal Ideation (SSI) | baseline, 6 weeks, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Treatment retention | 12 weeks
  Number of treatment sessions attended.

CONTACTS AND LOCATIONS:
Overall Officials: Guy S Diamond, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - CHOP Adolescent Care Center, Philadelphia, Pennsylvania
  - CHOP University City Primary Care, Philadelphia, Pennsylvania
  - CHOP Primary Care Center at Cobb's Creek, Philadelphia, Pennsylvania
  - CHOP Primary Care Center in South Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Diamond G, Creed T, Gillham J, Gallop R, Hamilton JL. Sexual trauma history does not moderate treatment outcome in Attachment-Based Family Therapy (ABFT) for adolescents with suicide ideation. J Fam Psychol. 2012 Aug;26(4):595-605. doi: 10.1037/a0028414. Epub 2012 Jun 18. PMID 22709259
- [Result] Diamond GS, Wintersteen MB, Brown GK, Diamond GM, Gallop R, Shelef K, Levy S. Attachment-based family therapy for adolescents with suicidal ideation: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2010 Feb;49(2):122-31. doi: 10.1097/00004583-201002000-00006. PMID 20215934